CLINICAL TRIAL: NCT02060630
Title: Best Endovascular Versus Best Surgical Therapy in Patients With Critical Limb Ischemia
Brief Title: Best Endovascular vs. Best Surgical Therapy in Patients With Critical Limb Ischemia
Acronym: BEST-CLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Boston Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Abbott (Industry); Bard Ltd (Industry); Boston Scientific Corporation (Industry); Cordis US Corp. (Industry); Abbott Medical Devices (Industry); Canadian Society for Vascular Surgery (Unknown); Eastern Vascular Society (Unknown); W.L.Gore & Associates (Industry); Midwest Vascular Society (Unknown); New England Society for Vascular Surgery (Unknown); Society for Clinical Vascular Surgery (Unknown); Society for Interventional Radiology (Unknown); Southern Vascular Society (Unknown); Society for Vascular Medicine (Unknown); Society for Vascular Surgery (Other); Vascular and Endovascular Surgery Society (Unknown); Vascular Interventional Advances (Unknown); Western Vascular Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEST-CLI Trial; 1U01HL107407 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2022-03

CONDITIONS: Critical Limb Ischemia
Keywords: Surgical revascularization; Endovascular revascularization; Amputation; Peripheral artery disease; Critical limb ischemia; claudication; leg pain; leg ulcer; gangrene
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Intermittent Claudication; Leg Ulcer; Gangrene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Available vein, open surg. revasc. (Other): Subjects with an available SSGSV cohort randomized to open surgical revascularization
  Interventions: Procedure: Open surgical revascularization
- Available vein, endovasc. revasc. (Other): Subjects with an available SSGSV cohort randomized to endovascular revascularization
  Interventions: Device: Endovascular revascularization
- Alternative conduit, open surg. revasc. (Other): Subjects with an alternative conduit cohort randomized to open surgical revascularization
  Interventions: Procedure: Open surgical revascularization
- Alternative conduit, endovasc. revasc. (Other): Subjects with an alternative conduit cohort randomized to endovascular revascularization
  Interventions: Device: Endovascular revascularization

INTERVENTIONS:
Procedure: Open surgical revascularization
  Arms: Alternative conduit, open surg. revasc.; Available vein, open surg. revasc.
Device: Endovascular revascularization — A variety of FDA approved devices will be used within this treatment arm. The trial will submit a proof-of-concept IDE application to the FDA to cover all devices.
  Arms: Alternative conduit, endovasc. revasc.; Available vein, endovasc. revasc.

SUMMARY:
This study will compare the effectiveness of best available surgical treatment with best available endovascular treatment in adults with critical limb ischemia (CLI) who are eligible for both treatment options.

DETAILED DESCRIPTION:
Male and female subjects aged 18 years or older will be randomized to receive either open surgical treatment or endovascular treatment. They will be followed for at least 2 years and up to 4 years and 2 months after treatment to primarily assess survival and major adverse limb events in the index or treated limb, and secondarily, to determine clinical and cost effectiveness outcomes after treatment. These outcomes (survival-free of major limb events and clinical, functional and cost effectiveness) will be compared within two cohorts of subjects: those with an available single-segment great saphenous vein, and those with an alternative conduit. The null hypotheses for both cohorts is that there will be no difference in MALE-free survival between best endovascular therapy and best surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older.
2. Infrainguinal PAOD (occlusive disease of the arteries below the inguinal ligament).
3. CLI, defined as arterial insufficiency with gangrene, non-healing ischemic ulcer, or rest pain consistent with Rutherford categories 4-6.
4. Candidate for both endovascular and open infrainguinal revascularization as judged by the treating investigators
5. Adequate aortoiliac inflow.
6. Adequate popliteal, tibial or pedal revascularization target defined as an infrainguinal arterial segment distal to the area of stenosis/occlusion which can support a distal anastomosis of a surgical bypass.
7. Willingness to comply with protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

1. Presence of a popliteal aneurysm (>2 cm) in the index limb.
2. Life expectancy of less than 2 years due to reasons other than PAOD.
3. Excessive risk for surgical bypass (as determined by the operating surgeon and the CLI Team)
4. Planned above ankle amputation on ipsilateral limb within 4 weeks of index procedure.
5. Active vasculitis, Buerger's disease, or acute limb-threatening ischemia
6. Any prior index limb infrainguinal stenting or stent grafting associated with significant restenosis within 1 cm of stent or stent-graft, unless the occlusion/restenosis site is outside the intended treatment zone (i.e.,. a tibial vessel that is not currently intended to be revascularized as a part of the treatment for CLI).
7. Any of the following procedures performed on the index limb within 3 months prior to enrollment:

   1. Infrainguinal balloon angioplasty, atherectomy, stent, or stentgraft;
   2. Infrainguinal bypass with either venous or prosthetic conduit
8. Open surgical inflow procedure (aortofemoral, axillofemoral, iliofemoral, thoracofemoral or femorofemoral bypass) within 6 weeks prior to enrollment
9. Current chemotherapy or radiation therapy.
10. Absolute contraindication to iodinated contrast due to prior near-fatal anaphylactoid reaction (laryngospasm, bronchospasm, cardiorespiratory collapse, or equivalent) which would preclude patient participation in angiographic procedures.
11. Pregnancy or lactation.
12. Administration of an investigational drug for PAD within 30 days of randomization.
13. Participation in a clinical trial (except observational studies) within the previous 30 days.
14. Prior enrollment or randomization into BEST-CLI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1843 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint: MALE (Major Adverse Limb Event)-free survival. MALE is defined as above ankle amputation of the index limb or major re-intervention (e.g. new bypass graft, jump/interposition graft revision, or thrombectomy/ thrombolysis) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  * Time to major adverse limb event or death, whichever occurs first in subjects with Single-Segment Great Saphenous Vein (SSGSV) available
  * Time to major adverse limb event or death, whichever occurs first in subjects without available SSGSV

SECONDARY OUTCOMES:
Clinical: Re-intervention and amputation-free survival (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention of the index leg, above ankle amputation of the index leg, or death, whichever occurs first in subjects with SSGSV available
Clinical: Re-intervention and amputation-free survival (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention of the index leg, above ankle amputation of the index leg, or death, whichever occurs first in subjects without available SSGSV
Clinical: Freedom from MALE-POD (POD, defined as death within 30 days of index procedure) (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention of the index leg, amputation of the index leg, or death within 30 days of index procedure, whichever occurs first in subjects with SSGSV available
Clinical: Clinical: Freedom from MALE-POD (POD, defined as death within 30 days of index procedure) (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention of the index leg, amputation of the index leg, or death within 30 days of index procedure, whichever occurs first in subjects without available SSGSV
Clinical: Amputation-free survival (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to amputation of the index leg, or death, whichever occurs first in subjects with SSGSV available
Clinical: Amputation-free survival (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to amputation of the index leg, or death, whichever occurs first in subjects without available SSGSV
Clinical: Freedom from POD (POD, defined as death within 30 days of index procedure) (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to death within 30 days of index procedure in subjects with SSGSV available
Clinical: Freedom POD (POD, defined as death within 30 days of index procedure) (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to death within 30 days of index procedure in subjects without available SSGSV
Clinical: Freedom from Myocardial Infarction (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to myocardial infarction (MI) in subjects with SSGSV available
Clinical: Freedom from Myocardial Infarction (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to myocardial infarction (MI) in subjects without available SSGSV
Clinical: Freedom from Stroke (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to stroke in subjects with SSGSV available
Clinical: Freedom from Stroke (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to stroke in subjects without available SSGSV
Clinical: Freedom from re-intervention (major and minor) in index leg (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention (major and minor) in index leg in subjects with SSGSV available
Clinical: Freedom from re-intervention (major and minor) in index leg (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to re-intervention (major and minor) in index leg in subjects without available SSGSV
Clinical: Number of re-interventions (major and minor) in per limb salvaged (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Number of re-interventions (major and minor) in per limb salvaged in subjects with SSGSV available
Clinical: Number of re-interventions (major and minor) in per limb salvaged (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Number of re-interventions (major and minor) in per limb salvaged in subjects without available SSGSV
Clinical: Freedom from hemodynamic failure (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to hemodynamic failure in subjects with SSGSV available
Clinical: Freedom from hemodynamic failure (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to hemodynamic failure in subjects without available SSGSV
Clinical: Freedom from clinical failure (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to above ankle amputation, major reintervention, MALE, degradation of WIfI stage or death, whichever occurs first in subjects with SSGSV available
Clinical: Freedom from clinical failure (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to above ankle amputation, major reintervention, MALE, degradation of WIfI stage or death, whichever occurs first in subjects without available SSGSV
Clinical: Freedom from Critical Limb Ischemia (CLI) (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to resolution of presenting CLI symptoms in the index limb in subjects with SSGSV available
Clinical: Freedom from Critical Limb Ischemia (CLI) (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to resolution of presenting CLI symptoms in the index limb in subjects without available SSGSV
Clinical: Freedom from all-cause mortality (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to all-cause mortality in subjects with SSGSV available
Clinical: Freedom from all-cause mortality (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Time to all-cause mortality in subjects without available SSGSV
Functional: Quality of Life assessment using VasuQoL (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  VasuQOL measurements in subjects with SSGSV available
Functional: Quality of Life assessment using VasuQoL (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  VasuQOL measurements in subjects without available SSGSV
Functional: Quality of Life assessment using EuroQoL (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  EuroQOL measurements in subjects with SSGSV available
Functional: Quality of Life assessment using EuroQoL (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  EuroQOL measurements in subjects without available SSGSV
Functional: Function assessment using SF-12, PCS (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Physical Component Summary (PCS) scores in subjects with SSGSV available
Functional: Function assessment using SF-12, PCS (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Physical Component Summary (PCS) scores in subjects without available SSGSV
Functional: Function assessment using SF-12, MCS (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Mental Component Summary (MCS) scores in subjects with SSGSV available
Functional: Function assessment using SF-12, MCS (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Mental Component Summary (MCS) scores in subjects without available SSGSV
Functional: Function assessment using SF-12, SF-6D R2 (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Utility Index (SF-6D R2) scores in subjects with SSGSV available
Functional: Function assessment using SF-12, SF-6D R2(cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Utility Index (SF-6D R2) scores in subjects without available SSGSV
Functional: Numerical rating scale for Pain, Pain Now (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Pain Now in subjects with SSGSV available
Functional: Numerical rating scale for Pain, Pain Now (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Pain Now in subjects without available SSGSV
Functional: Numerical rating scale for Pain, Usual level of Pain (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Usual level of Pain during the last week in subjects with SSGSV available
Functional: Numerical rating scale for Pain, Usual level of Pain (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Usual level of Pain during the last week in subjects without available SSGSV
Functional: Numerical rating scale for Pain, Best level of Pain (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Best level of Pain during the last week in subjects with SSGSV available
Functional: Numerical rating scale for Pain, Best level of Pain (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Best level of Pain during the last week in subjects without available SSGSV
Functional: Numerical rating scale for Pain, Worst level of Pain (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Worst level of Pain during the last week in subjects with SSGSV available
Functional: Numerical rating scale for Pain, Worst level of Pain (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Scores for Worst level of Pain during the last week in subjects without available SSGSV
Function: Six-minute walk test (cohort 1) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Six-minute walk test measurements in subjects with SSGSV available. The six-minute walk test was performed at a subset of clinical sites (for whom this test was standard of care) and was limited to patients for whom rest pain, wounds, or foot surgery (recent or anticipated) did not preclude weight bearing
Function: Six-minute walk test (cohort 2) | Through each subject's last regularly scheduled study visit, up to a maximum of 84 months per subject
  Six-minute walk test measurements in subjects without available SSGSV. The six-minute walk test was performed at a subset of clinical sites (for whom this test was standard of care) and was limited to patients for whom rest pain, wounds, or foot surgery (recent or anticipated) did not preclude weight bearing

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Menard, MD, Principal Investigator — Brigham and Women's Hospital; Alik Farber, MD, Principal Investigator — Boston University; Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Mark Cziraky, PharmD, CLS, Principal Investigator — Carelon Research; Taye Hamza, PhD, Principal Investigator — Carelon Research
Locations (161):
- United States (144):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Heart Hospital, Phoenix, Arizona
  - University of Arizona - Banner University Medical Center, Tucson, Arizona
  - Carondelet Heart & Vascular Institute, Tucson, Arizona
  - University of Arkansas for Medical Services, Little Rock, Arkansas
  - University of California - Irvine, Irvine, California
  - San Diego VAMC, La Jolla, California
  - UC San Diego Sulpizio Cardiovascular Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda VA Medical Center, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - VA Greater Los Angeles, Los Angeles, California
  - Keck Medical Center of USC, Los Angeles, California
  - UCLA-Gonda Vascular Surgery, Los Angeles, California
  - VA Palo Alto Health Care, Palo Alto, California
  - Sacramento VA Medical Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente (San Diego), San Diego, California
  - Kaiser Permanente Northern California, San Francisco, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California-San Francisco Medical Center, San Francisco, California
  - Stanford Hospital, Stanford, California
  - Harbor - UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health, Denver, Colorado
  - Vascular Institute of the Rockies, Denver, Colorado
  - Rocky Mountain Regional VA, Denver, Colorado
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - West Haven VAMC, West Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - GW Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - University of Florida (Gainesville), Gainesville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Miami, Miami Springs, Florida
  - Florida Hospital Ocala, Ocala, Florida
  - Tampa General Hospital, Tampa, Florida
  - Tampa VAMC, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Kaiser Foundation Hospital, Honolulu, Hawaii
  - Central DuPage Hospital (Cadence), Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Memorial Hospital, Winfield, Illinois
  - Indiana University Medical School, Indianapolis, Indiana
  - Mercy Hospital Medical Center, West Des Moines, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - University Health System: LSU Health Sciences, Shreveport, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Loyola University Medical Center, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Steward St. Elizabeth's Medical Center, Brighton, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Michigan Heart/St. Joseph Mercy Ann Arbor Hospital, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Hospital/Abbott Northwestern Hosp., Minneapolis, Minnesota
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Midwest Aortic Vascular Institute, Kansas City, Missouri
  - St. Louis VA Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Hanover, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New Mexico VA Medical Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - VA Western NY Healthcare System, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Vascular Health Partners, Queensbury, New York
  - University of Rochester Medical Center, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook Medicine, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Durham VAMC, Durham, North Carolina
  - North Carolina Heart and Vascular Research, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals of Cleveland/Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Oklahoma College of Medicine at Tulsa, Tulsa, Oklahoma
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health System, Wormleysburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital/Brown Medical School, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health-Upstate (Formerly Greenville Memorial Hospital), Greenville, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Memorial Hermann Hospital TMC, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Scott and White - Temple, Temple, Texas
  - The University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Meriter Wisconsin Heart, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Milwaukee VAMC, Milwaukee, Wisconsin
- Canada (12):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - University of Western Ontario, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill, Montreal, Quebec
  - Jewish General Hostpital, Montreal, Quebec
  - Chu de Quebec, Québec, Quebec
  - Regina Qu'Appelle, Regina, Saskatchewan
  - St. Paul's Hospital, Saskatoon, Saskatchewan
- Helsinki University Hospital, Helsinki, Finland
- San Giovanni di Dio Hospital, Florence, Italy
- New Zealand (3):
  - Auckland City Hospital, Grafton, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
  - Wellington Hospital, Newtown, Wellington Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hicks CW, Farber A, Doros G, Kinlay S, Powell RJ, Strong MB, Rosenfield K, Aridi H, Motaganahalli R, Barleben A, Siracuse JJ, Azene E, Malas M, Conte MS, Zayed M, Menard MT. Atherectomy Is Not Associated With Improved Limb-Based Outcomes Among Patients in the BEST-CLI Trial Undergoing Endovascular Revascularization. JACC Cardiovasc Interv. 2026 Jan 12;19(1):96-107. doi: 10.1016/j.jcin.2025.10.065. PMID 41534992
- [Derived] Venermo MA, de Vega M, Houlind K, Siracuse JJ, Doros G, Kiang S, Barshes N, Rosenfield K, Menard MT, Farber A; BEST-CLI hemodynamic working group. Baseline Haemodynamic Measurements and Immediate Change in Parameters after Revascularisation: Ankle Pressure, Ankle Brachial Index, Toe Pressure, and Toe Brachial Index Analysis of the BEST-CLI Participants. Eur J Vasc Endovasc Surg. 2025 Dec 24:S1078-5884(25)01311-5. doi: 10.1016/j.ejvs.2025.12.042. Online ahead of print. PMID 41453560
- [Derived] Conte MS, Farber A, Barleben A, Chisci E, Doros G, Kashyap VS, Kayssi A, Kolh P, Moreira CC, Nypaver T, Rosenfield K, Rowe VL, Schanzer A, Singh N, Siracuse JJ, Strong MB, Menard MT. Impact of Bypass Conduit and Early Technical Failure on Revascularization for Chronic Limb-Threatening Ischemia. Circ Cardiovasc Interv. 2025 Mar;18(3):e014716. doi: 10.1161/CIRCINTERVENTIONS.124.014716. Epub 2025 Mar 18. PMID 40100950
- [Derived] Siracuse JJ, Farber A, Menard MT, Conte MS, Kaufman JA, Jaff M, Kiang SC, Ochoa Chaar CI, Osborne N, Singh N, Tan TW, Guzman RJ, Strong MB, Hamza TH, Doros G, Rosenfield K. Perioperative complications following open or endovascular revascularization for chronic limb-threatening ischemia in the BEST-CLI Trial. J Vasc Surg. 2023 Oct;78(4):1012-1020.e2. doi: 10.1016/j.jvs.2023.05.040. Epub 2023 Jun 14. PMID 37318428
- [Derived] Levin SR, Farber A, Kobzeva-Herzog A, King EG, Eslami MH, Garg K, Patel VI, Rockman CB, Rybin D, Siracuse JJ. Postoperative disability and one-year outcomes for patients suffering a stroke after carotid endarterectomy. J Vasc Surg. 2023 Aug;78(2):413-422.e1. doi: 10.1016/j.jvs.2023.04.002. Epub 2023 Apr 10. PMID 37040850
- [Derived] Siracuse JJ, Rowe VL, Menard MT, Rosenfield K, Conte MS, Powell R, Clavijo LC, Giles KA, Hamza TH, Van Over M, Cziraky M, White CJ, Strong MB, Farber A. Relationship between WIfI stage and quality of life at revascularization in the BEST-CLI trial. J Vasc Surg. 2023 Apr;77(4):1099-1106.e4. doi: 10.1016/j.jvs.2022.11.050. Epub 2022 Nov 23. PMID 36435274
- [Derived] Farber A, Menard MT, Conte MS, Kaufman JA, Powell RJ, Choudhry NK, Hamza TH, Assmann SF, Creager MA, Cziraky MJ, Dake MD, Jaff MR, Reid D, Siami FS, Sopko G, White CJ, van Over M, Strong MB, Villarreal MF, McKean M, Azene E, Azarbal A, Barleben A, Chew DK, Clavijo LC, Douville Y, Findeiss L, Garg N, Gasper W, Giles KA, Goodney PP, Hawkins BM, Herman CR, Kalish JA, Koopmann MC, Laskowski IA, Mena-Hurtado C, Motaganahalli R, Rowe VL, Schanzer A, Schneider PA, Siracuse JJ, Venermo M, Rosenfield K; BEST-CLI Investigators. Surgery or Endovascular Therapy for Chronic Limb-Threatening Ischemia. N Engl J Med. 2022 Dec 22;387(25):2305-2316. doi: 10.1056/NEJMoa2207899. Epub 2022 Nov 7. PMID 36342173
- [Derived] Albaghdadi MS, Young MN, Chowdhury MM, Assmann S, Hamza T, Siami S, Villarreal M, Strong M, Menard M, Farber A, Rosenfield K. Clinical practice patterns and ascertainment bias for cardiovascular events in a randomized trial: A survey of investigators in the BEST-CLI trial. Vasc Med. 2021 Apr;26(2):180-186. doi: 10.1177/1358863X21995897. PMID 33825577
- [Derived] Rathakrishnan B, Secemsky EA. Turning the tide: Evolution of below-the-knee endovascular intervention. Vasc Med. 2021 Feb;26(1):26-27. doi: 10.1177/1358863X20978281. Epub 2020 Dec 14. No abstract available. PMID 33314979
- [Derived] Powell R, Menard M, Farber A, Rosenfield K, Goodney P, Gray B, Lookstein R, Pena C, Schermerhorn M. Comparison of specialties participating in the BEST-CLI trial to specialists treating peripheral arterial disease nationally. J Vasc Surg. 2019 May;69(5):1505-1509. doi: 10.1016/j.jvs.2018.08.188. PMID 31010516
- [Derived] Farber A, Rosenfield K, Siami FS, Strong M, Menard M. The BEST-CLI trial is nearing the finish line and promises to be worth the wait. J Vasc Surg. 2019 Feb;69(2):470-481.e2. doi: 10.1016/j.jvs.2018.05.255. PMID 30683195
- [Derived] Menard MT, Farber A, Assmann SF, Choudhry NK, Conte MS, Creager MA, Dake MD, Jaff MR, Kaufman JA, Powell RJ, Reid DM, Siami FS, Sopko G, White CJ, Rosenfield K. Design and Rationale of the Best Endovascular Versus Best Surgical Therapy for Patients With Critical Limb Ischemia (BEST-CLI) Trial. J Am Heart Assoc. 2016 Jul 8;5(7):e003219. doi: 10.1161/JAHA.116.003219. PMID 27402237